CLINICAL TRIAL: NCT05205941
Title: A Phase 1b Study to Assess the Safety, Tolerability and Antimalarial Activity of MMV533 Against Plasmodium Falciparum Blood Stage Infection in Healthy Volunteers
Brief Title: MMV533 Plasmodium Falciparum Volunteer Infection Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Nucleus Network Ltd (Other); Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MMV_MMV533_20_01
Record Dates: First submitted 2021-08-31; First posted 2022-01-25 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Malaria
Keywords: Tolerability; Safety
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MMV533 (single, oral doses). (Other): Approximately 12 volunteers in 1 cohort, Up to six dose levels between 10 and 160mg
  Interventions: Drug: MMV688533

INTERVENTIONS:
Drug: MMV688533 — Not exceeding 200mg
  Other Names: MMV533

SUMMARY:
A Phase 1b study to assess the safety, tolerability and antimalarial activity of MMV533 against Plasmodium falciparum 3D7 blood stage infection in healthy volunteers

DETAILED DESCRIPTION:
The study will characterise the effects of single oral doses of MMV533 on the clearance of Plasmodium falciparum 3D7 using the Induced Blood Stage Malaria (IBSM) model. This is a well-established method for obtaining useful pharmacokinetic-pharmacodynamic (PK-PD) information on anti-malarial drugs.

The study will be an open-label, pilot Volunteer Infection Study (VIS) using the IBSM model and single dose IMP. The study will be conducted in healthy malaria-naive adult volunteers infected with Plasmodium falciparum 3D7, in one cohort of approximately 12 volunteers (all receiving active treatment). From an operational perspective, the full cohort may be conducted in subgroups of up to 6 volunteers. Ascending doses will be administered in order of enrolment number (per sub-group, if applicable). Volunteers will be enrolled within a 28 day screening period to ensure volunteers meet all the inclusion criteria and none of the exclusion criteria.

On Day -8 (8 days prior to IMP administration), volunteers will attend the clinical unit to be inoculated with the malaria challenge agent containing approximately 2,800 viable human erythrocytes infected with P. falciparum 3D7 parasites. Parasitaemia will be monitored on an outpatient basis daily on Day -4, and then twice daily on Day -3, Day -2 and until admission to the clinical unit on Day -1 for eligibility check and confinement.

Volunteers will be administered IMP on Day 1 and will have safety monitoring and blood sampling for parasitaemia monitoring and PK analysis on an inpatient basis for at least 108 hours post-IMP administration. Volunteers will be discharged from the clinical unit after review of ECG, vital signs, clinical and laboratory tests safety data by the Principal Investigator or delegate, and will then attend the clinical unit on an outpatient basis regularly for continued safety monitoring and blood sampling for parasitaemia monitoring and PK analysis.

Volunteers will be administered mandatory malaria rescue medication at Day 21±3, or earlier if there is failure to clear parasites or recrudescence and at the discretion of the Principal Investigator or delegate. EOS will be on Day 28±3. Volunteers must have had at least two negative 18S qPCR (18 Svedberg quantitative polymerase chain reaction) results prior to EOS and must have completed their course of anti-malarial rescue medication.

In the event of recrudescence, blood samples will be collected prior to rescue treatment to culture parasites for drug resistance testing.

ELIGIBILITY:
Inclusion Criteria:

1. Having given written informed consent prior to undertaking any study-related procedure.
2. Male or female aged between 18 to 55 years inclusive.
3. Available for the duration of the study and for 2 weeks following the End of Study Visit (EOS).
4. Lives with a spouse, family member, or housemate from the time of inoculation with the malaria challenge agent through to the EOS.
5. Total body weight greater than or equal to 50 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive).
6. Willing to defer blood donations to a blood service for a minimum of 6 months after the EOS.
7. Heterosexual women of childbearing potential (WOCBP) must agree to the use of a highly effective method of birth control (see below) combined with a barrier contraceptive from the screening visit until 30 days after the last dose of the IMP (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of IMP) and have a negative result on urine pregnancy test performed before inoculation with the malaria challenge agent.
8. Women of non-childbearing potential (WONCBP)
9. Males who have, or may have female sexual partners of child bearing potential during the course of the study must agree to use a double method of contraception including condom plus diaphragm, or condom plus intrauterine device, or condom plus stable oral/transdermal/injectable/implantable hormonal contraceptive by the female partner, from the time of informed consent through to 60 days (covering a spermatogenesis cycle) after the last dose of the IMP. Abstinent males must agree to start a double method if they begin sexual relationship with a female during the study and up to 60 days after the last dose of study drug. Males with female partners of child-bearing potential that are surgically sterile, or males who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception.
10. Vital signs after 5 minutes resting in supine position:

    1. Systolic blood pressure (SBP) - 90-140 mmHg,
    2. Diastolic blood pressure (DBP) - 40-90 mmHg,
    3. Heart rate (HR) 40-100 bpm.

At Screening and pre-inoculation with the malaria challenge agent: normal standard mean of triplicate 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges:

1. QT ≤ 500 msec,
2. QT Interval Corrected Using Fridericia's Formula (QTcF) QTcF ≤ 450 msec, QT Interval Corrected Using Bazett's Formula (QTcB) QTcB ≤ 450 msec
3. PR interval ≤ 210 msec for both males and females, and
4. Normal ECG tracing unless the Principal Investigator or delegate considers an ECG tracing abnormality to be not clinically relevant.

   12. In the opinion of the Principal Investigator or delegate, the individual has a high probability of adherence with and completion of the study, and willing and able to withdraw and refrain from restricted medications.

   13. Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

   14. Fluent in English and able to understand and comply with written and verbal protocol-related requirements.

   15. Agrees to adhere to the lifestyle considerations throughout the study (see Section 4.3.3) and is willing to consume 240 mL full-fat milk with each dose of rescue medication Riamet®.

   Exclusion Criteria:
   1. Any lifetime history of malaria or participation in a previous malaria challenge study or malaria vaccine trial.
   2. Must not have had malaria exposure that is considered significant by the Principal Investigator or delegate. This includes but is not limited to:

      * history of having travelled to or lived (> 2 weeks) in a malaria-endemic region during the past 12 months or planned travel to a malaria-endemic region during the course of the trial;
      * history of having lived for >1 year in a malaria-endemic region in the past 10 years;
      * history of having ever lived in a malaria-endemic region for more than 10 years inclusive. For endemic regions see https://malariaatlas.org/explorer/#/ Bali is not considered a malaria-endemic region.
   3. Presence of acute infectious disease and/or abnormal body temperature (defined as an a.m. tympanic temperature >37.5 ºC or a p.m. >37.7 ºC) at pre-inoculation.
   4. Haematology, biochemistry or urinalysis results that are outside of the laboratory normal reference ranges and are either:

      * considered clinically significant by the Principal Investigator or delegate; OR
      * considered not clinically significant by the Principal Investigator or delegate but are also outside of Sponsor-approved clinically acceptable laboratory ranges
   5. Breastfeeding or lactating; positive serum pregnancy test at screening, positive urine pregnancy test upon admission or at other timepoints as specified by schedule of activities tables.
   6. Has previously received a blood transfusion.
   7. Use of antibiotics within 6 weeks of Screening.
   8. Use of systemic therapies with antimalarial activity within 6 weeks of Screening. This includes (but not limited to) artemisinin, amodiaquine, atovaquone, chloroquine, mefloquine, mepacrine, primaquine, proguanil, quinine, sulfadoxine-pyrimethamine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, doxycycline, and tafenoquine.
   9. Prior to screening and inoculation with the malaria challenge agent:

      * any systemic administration (oral, pulmonary/nasal, IV) of corticosteroids, anti-inflammatory drugs (excluding commonly used over-the-counter anti-inflammatory drugs such as ibuprofen, acetylsalicylic acid, diclofenac), immunomodulators or anticoagulants within the past three months.
      * Ibuprofen (preferred) may be used at doses of up to 1.2 g/day, or paracetamol at doses of up to 2 g/day after discussion with the Investigator. Limited use of other non-prescription medications or dietary supplements, not believed to affect subject safety or the overall results of the study, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the Investigator.
      * Any topical administration (cutaneous, eye drops) of corticosteroids within the past 2 weeks.
      * Any individual currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration potentially associated with hypothalamic-pituitary-adrenal axis suppression within the past 12 months.
   10. Any contra-indication to rescue medication according to the applicable labelling and if found to be severely glucose-6-phosphate dehydrogenase (G6PD) deficient at screening (i.e. activity of less than 10% as per World Health Organization (WHO) definition).
   11. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic/ gallbladder*/ bile duct, renal, metabolic, haematological, neurological, musculoskeletal, rheumatologic, systemic, ocular, gynaecologic (if female), infectious or autoimmune disease, or signs of acute illness. *including medical history of asymptomatic gallbladder stones.
   12. History of recurrent headache (eg, tension-type, cluster or migraine) with a frequency of ≥2 episodes per month on average and severe enough to require medical therapy. History of recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
   13. Asthma (excluding childhood asthma, or mild asthma with preventative asthma medication required less than monthly and no event requiring treatment in the last 2 weeks prior to screening).
   14. Any personal history of surgical procedures that may affect IMP absorption, distribution (i.e. GI surgery) and metabolism or immune response to malaria inoculation (splenectomy).
   15. Blood donation of any volume within one month before screening, or participation in any research study involving blood sampling (more than 450 mL/unit of blood).
   16. Any documented evidence of current or past cardiovascular disease including:

       * cardiac arrhythmias or
       * family history of congenital long QT syndrome, Brugada syndrome, or unexplained sudden cardiac death.
       * Symptomatic postural hypotension at screening irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 3 min when changing from supine to standing position.
   17. Has evidence of increased cardiovascular risk (defined as >10%, 5-year risk for those greater than 35 years of age, as determined by the Australian Absolute Cardiovascular Disease Risk Calculator (http://www.cvdcheck.org.au). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, total and High-density lipoprotein (HDL) cholesterol (mmol/L) and reported diabetes status. Note: The site investigator will perform cardiovascular risk calculation once all assessments have been performed, prior to eligibility.
   18. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies, or any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Individuals with known lactose or dairy intolerance are excluded. Volunteers with seasonal allergies/hay fever or allergy to animals or house dust mite that are untreated and asymptomatic at the time of dosing can be enrolled in the trial.
   19. History of convulsion (including drug or vaccine-induced episodes). A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
   20. History of substance use disorder(s) within 5 years of screening and/or history of alcohol dependancy and/or any prior intravenous use of an illicit substance.
   21. Smoked > 1 pack of cigarettes per day for > 10 years, or who currently (within 14 days prior to screening) smokes > 5 cigarettes per day.
   22. Any individual who, in the judgement of the Principal Investigator or delegate, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
   23. Any individual who cannot be contacted in case of emergency.
   24. Any individual who is the Investigator, or delegates, research assistant, pharmacist, study coordinator, project manager, or other staff thereof, directly involved in conducting the study.
   25. Any individual without a good peripheral venous access.
   26. Participation in any investigational product study within the 12 weeks preceding inoculation with the malaria challenge agent or 5 times the half-life of the Investigational product, whichever is longer.
   27. Positive serology test for hepatitis B (HB) (positive Hepatitis B surface antigen (HB sAG) or anti-hepatitis B core antibody (anti-HBc Ab), hepatitis C (anti-HCV) or human immune deficiency virus (HIV) (positive for anti-HIV1 (HIV type 1) and anti-HIV2 (HIV type 2) Ab ).
   28. Positive urine drug test at Screening, prior to inoculation with the malaria challenge agent or prior to IMP dosing. Any drug from the list of drugs tested (such as amphetamine, barbiturates, benzodiazepines, cocaine, methamphetamine, methadone, Opiates, phencyclidine, Tetrahydrocannabinol; and their metabolites) unless there is an acceptable explanation to the Principal Investigator or delegate (eg, volunteer has stated in advance that they consumed a prescription of over the counter product which contained the detected drug) and/or the volunteer has a negative urine drug screen on retest.
   29. Positive alcohol screen at Screening, prior to inoculation with the malaria challenge agent or prior to IMP dosing.
   30. Any consumption of citrus fruits (such as grapefruit, Seville oranges) or their juices within 7 days prior to IMP administration.
   31. History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to: past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening.
   32. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer considered treated and cured), treated or untreated, within 5 years of Screening, regardless of whether there is no evidence of local recurrence or metastases.
   33. Any vaccination within 28 days of screening.
   34. Any medical condition that in the opinion of the Principal Investigator or delegate would jeopardize the individual's involvement in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Brisbane Clinic, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bestgen B, Jones S, Thathy V, Kuemmerle A, Barcelo C, Haouala A, Gossen D, Marx MW, Di Resta I, Szramowska M, Webster RA, Llewellyn S, Ritacco DA, Yeo T, Leroy D, Barber BE, Fidock DA, Griffin P, Lickliter J, Chalon S. Safety, tolerability, pharmacokinetics, and antimalarial activity of MMV533: a phase 1a first-in-human, randomised, ascending dose and food effect study, and a phase 1b Plasmodium falciparum volunteer infection study. Lancet Infect Dis. 2025 May;25(5):507-518. doi: 10.1016/S1473-3099(24)00664-9. Epub 2024 Dec 18. PMID 39708824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nine (9) participants were inoculated with the malaria challenge agent, 7 of whom were subsequently administered 20 mg MMV533 (n=3), 35 mg (n=2) and 100 mg (n=2) MMV533.
  2 participants were not inoculated.
Groups:
- MMV533 (20 mg).: MMV 533 (20 mg) - (N=3 participants)
- MMV 533 (35 mg): MMV 533 (35 mg) - (N=2 participants)
- MMV533 (100 mg): MMV 533 (100 mg) (N=2 participants)
- Not Treated: Not treated - (N=2 participants)
Period: Overall Study
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg) | Not Treated
Started | 3 | 2 | 2 | 2
Completed | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MMV533 20 mg: Participants having been dosed with MMV533 20mg
- MMV533 35 mg: Participants having been dosed with MMV533 35mg
- MMV533 100 mg: Participants having been dosed with MMV533 100mg
- Not Treated: Participants not having been dosed with MMV533
- Total: Total of all reporting groups
Arm/Group | MMV533 20 mg | MMV533 35 mg | MMV533 100 mg | Not Treated | Total
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 9
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 32 (13.1) | 24.5 (7.8) | 22 (4.2) | 22.5 (2.1) | 26 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 2 | 1 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 2 | 1 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 2 | 2 | 2 | 9
BMI (kg/m2)* [Mean (Standard Deviation); unit: kg/m2] | 24.17 (1.91) | 23.55 (1.2) | 22.45 (2.19) | 27.25 (4.31) | 24.33 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: The Activity of Single Oral Doses of MMV533 (Name of Investigational Medicinal Product) on Clearance of Plasmodium
Description: Estimated Parasite Reduction Ratio over 48 hours (PRR48)
Time Frame: 48 hours
Measure: Geometric Mean (95% Confidence Interval); unit: PRR48=parasite reduction ratio 48 hours
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
PRR48=parasite reduction ratio 48 hours | 42.17 [20.23 to 87.90] | 158.03 [93.62 to 266.75] | 187.57 [96.72 to 363.77]

2. Primary Outcome: The Activity of Single Oral Doses of MMV533 (Name of Investigational Medicinal Product) on Clearance of Plasmodium
Description: Estimated Parasite Reduction Ratio over 48 hours (log10 PRR48)
Time Frame: 48 hours
Measure: Geometric Mean (95% Confidence Interval); unit: Log10 PRR48
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Log10 PRR48 | 1.62 [1.31 to 1.94] | 2.2 [1.97 to 2.43] | 2.27 [1.99 to 2.56]

3. Primary Outcome: The Activity of Single Oral Doses of MMV533 (Name of Investigational Medicinal Product) on Clearance of Plasmodium
Description: Parasite Clearance Half-life after Single Oral Dose of MMV533, by Treatment Group
Time Frame: 48 hours
Population: All participants (n=7) had significant regression models at the p=0.001 significance level and all contributed towards the dose specific PRR48 calculated.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Hours | 8.89 [7.43 to 11.06] | 6.57 [5.96 to 7.33] | 6.36 [5.64 to 7.28]

4. Primary Outcome: Participants With Parasitaemia Below Limit of Quantification (LOQ)
Description: Number of volunteers whose parasitaemia levels fall below limit of quantification (LOQ) following treatment with IMP
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Participants | 1 | 2 | 2

5. Primary Outcome: Activity of Single Oral Doses of MMV533 on Clearance of Plasmodium
Description: The Total Number of Study Participants with Recrudescence of Asexual Parasitaemia within 30 days post inoculation
Time Frame: 30 days post inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Participants | 0 | 2 | 0

6. Primary Outcome: The Activity of Single Oral Doses of MMV533 on Clearance of Plasmodium
Description: Number of participants experiencing a recrudescence after 180 hours
Time Frame: 180 hours post inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Participants | 0 | 1 | 0

7. Primary Outcome: The Activity of Single Oral Doses of MMV533 on Clearance of Plasmodium
Description: Number of participants experiencing a recrudescence after 312 hours
Time Frame: 312 hours post inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | MMV533 (20 mg). | MMV 533 (35 mg) | MMV533 (100 mg)
Number analyzed (Participants) | 3 | 2 | 2
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported up to 28 days from the time of inoculation with the malaria challenge agent . Medically untoward events between time of consent and inoculation with the malaria challenge agent were reported as medical history and not AEs.
Groups:
- MMV533 20mg (Single, Oral Doses): MMV533 20mg
- MMV533 35mg (Single, Oral Doses): MMV533 35mg
- MMV533 100mg (Single, Oral Doses): MMV533 100mg
Arm/Group | MMV533 20mg (Single, Oral Doses) | MMV533 35mg (Single, Oral Doses) | MMV533 100mg (Single, Oral Doses)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT05205941/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT05205941/SAP_001.pdf
  • Informed Consent Form (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT05205941/ICF_002.pdf